CLINICAL TRIAL: NCT01688817
Title: The Magnitude of Effect of Physician's Counseling on Participation Rate and Utilization of Sedation in Colonoscopy-based Colorectal Cancer Screening Program
Brief Title: The Magnitude of Effect of PCP Counseling on Participation Rate and Sedation Rate in Colonoscopy-based Screening Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMKP-2008
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Colonoscopy; Early Detection of Cancer; Patient Selection; Patient Participation; Physicians, Primary Care; Conscious Sedation
MeSH Terms: conditions — Colorectal Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician's counseling (Other)
  Interventions: Other: Physician's counseling
- Information leaflet (Active Comparator)
  Interventions: Other: Information leaflet

INTERVENTIONS:
Other: Physician's counseling — Colorectal cancer (CRC) screening was recommended to a patient personally by a PCP. The issue was discussed during a routine medical visit according to a standardized scheme. PCP provided a patient with a rationale for CRC screening in asymptomatic individuals and benefits of early treatment of the disease. A patient was told about colonoscopy-based screening program. A PCP provided patient with information on how colonoscopy is performed and how to prepare a bowel for the examination, and informed a patient about possible adverse events related to the procedure including post-polypectomy bleeding and bowel perforation. According to the scheme of the discussion screening modalities other than colonoscopy were not debated, unless a patient specifically asked about them.
  Arms: Physician's counseling
Other: Information leaflet — Patients were given leaflet on primary colonoscopy colorectal cancer screening program. A leaflet provided rationale for colorectal cancer screening and information on colonoscopy-based colorectal cancer screening program.
  Arms: Information leaflet

SUMMARY:
The purpose of this study is to assess the impact of physician's counseling on participation and utilization of sedation in a primary colonoscopy-based colorectal cancer (CRC) screening program

DETAILED DESCRIPTION:
Participation rate is one of the major factors influencing the effectiveness of screening programs. Participation rates in CRC screening, including primary colonoscopy programs, remain suboptimal. It is known that one of the strongest predictors of CRC screening participation rate is a physician, especially primary care physician (PCP), recommendation. Engaging a PCP tends to improve participation rate in organized and opportunistic cancer screening programs.

To our best knowledge there are no randomized controlled trials, dedicated specifically to assess the effect of physician's counseling on participation rate in primary colonoscopy CRC screening programs. There is also no data on the impact of physician's counseling on patient's decision to choose unsedated (not in sedation) or sedated colonoscopy.

In this study we aimed to quantitatively estimate the impact of a PCP's counseling on screening participation rate and utilization of sedation in the opportunistic primary CRC screening program when compared to the effect obtained by using a standardized information leaflet only.

ELIGIBILITY:
Inclusion Criteria:

* 50-65 years of age

Exclusion Criteria:

* colonoscopy within last 10 years
* change in bowel habits in the previous six months
* a visible blood in stool (unless related to known hemorrhoids)
* anemia or weight loss of unknown cause
* severe comorbid conditions making subject ineligible for screening colonoscopy

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Effect of primary care physician's (PCP) counseling on participation rate in primary colonoscopy screening program | Six months after intervention

SECONDARY OUTCOMES:
Effect of primary care physician's (PCP) counseling on a patient's decision to choose unsedated colonoscopy (not in sedation). | Six months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Regula, MD, PhD, Study Director — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology; Michal F. Kaminski, MD, PhD, Study Chair — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland; Michal Wiszniewski, MD, Principal Investigator — The Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland

REFERENCES:
- [Derived] Boguradzka A, Wiszniewski M, Kaminski MF, Kraszewska E, Mazurczak-Pluta T, Rzewuska D, Ptasinski A, Regula J. The effect of primary care physician counseling on participation rate and use of sedation in colonoscopy-based colorectal cancer screening program--a randomized controlled study. Scand J Gastroenterol. 2014 Jul;49(7):878-84. doi: 10.3109/00365521.2014.913191. Epub 2014 May 5. PMID 24797871